CLINICAL TRIAL: NCT02183194
Title: A Prospective, MultiCenter, Single-arm, Post-market Study of Paclitaxel Coated PTA Balloons for Treatment of Dysfunctional AV Fistulae and Grafts (ACCESS)
Brief Title: Paclitaxel Coated PTA Balloons for Treatment of Dysfunctional AV Fistulae and Grafts
Acronym: ACCESS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0021-01
Record Dates: First submitted 2014-06-25; First posted 2014-07-08 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Dysfunctional AV Graft; Dysfunctional AV Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lutonix Paclitaxel Drug Coated Balloon (Experimental)
  Interventions: Device: Lutonix Paclitaxel Drug Coated Balloon

INTERVENTIONS:
Device: Lutonix Paclitaxel Drug Coated Balloon

SUMMARY:
The purpose of this study is to evaluate the Lutonix® 035 Drug Coated Balloon PTA Catheter (CE mark) for use as intended in the treatment of subjects with clinically significant hemodialysis vascular access stenosis or occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the informed consent form (ICF)
3. Hemodialysis access on the arm presenting with any clinical abnormalities as defined in the K/DOQI guidelines
4. Native AV fistula or synthetic AV graft has been implanted ≥30 days
5. Target de novo or non-stented restenotic lesion(s) consisting of a >50% stenosis by visual estimate. Successful treatment of non target lesion(s) (residual stenosis <30% by visual estimate) without procedural complication by standard of care
6. Successful predilatation of the target lesion with a percutaneous transluminal angioplasty (PTA) balloon
7. Intended target lesion(s) (maximum of 2) can be treated
8. No other prior surgical or vascular interventions within 2 weeks before and/or planned 30 days after the treatment

Exclusion Criteria:

1. Women who are pregnant, lactating, or planning on becoming pregnant or men intending to father children
2. Known contraindication (including allergic reaction) or sensitivity to contrast media, ASA, clopidogrel, ticlopidine, paclitaxel (mild to severe cases), that cannot be adequately managed with pre-and post-procedure medication
3. Life expectancy <12months
4. Scheduled for kidney transplant or peritoneal dialysis in the next 12months;
5. Thrombosed access
6. Stent in the target treatment area
7. Blood coagulative disorder, sepsis, or current AV access infection
8. Currently participating in an investigational drug, biologic, or device study, or previous enrollment in this study NOTE: Enrollment in another investigational drug, biologic, or device study during the follow- up period is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: Primary Patency | 6 months
  Target Lesion Primary Patency (TLPP): The interval following index procedure intervention until the next reintervention of the target lesion or access thrombosis.

SECONDARY OUTCOMES:
Target Lesion Primary Patency (TLPP) | 12 months
Access circuit primary patency | 6 and 12 months
Abandonment of permanent access in the index extremity | 6 and 12 months
Number of interventions required to maintain target lesion patency | 6 and 12 months
Number of interventions, required to maintain access circuit patency | 6 and 12 months
  The access circuit is defined as "the area from the AV access graft arterial anastomosis to the superior vena-cava right atrial junction." The outcome is recording all interventions that occur in the access circuit up until the time of circuit failure (patency).
Major vascular complications | < or at 1 month
Rate of device and procedure related adverse events | 1, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Austria (2):
  - LKH-Univ. Klinikum Graz, Graz
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
- Germany (2):
  - Universitätsklinikum Köln AöR, Cologne
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck